CLINICAL TRIAL: NCT05172843
Title: Comparison of Intensive Diet With Knee Arthroplasty for Treatment of Obese Patients With Knee Osteoarthritis: a Randomized Trial
Brief Title: Intensive Diet vs Knee Arthroplasty for Knee Osteoarthritis
Acronym: INKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marius Henriksen (Other)
Responsible Party: Sponsor-Investigator, Marius Henriksen, Professor, Frederiksberg University Hospital
Organization: Frederiksberg University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: APPI2-OA-2021-01
Record Dates: First submitted 2021-12-13; First posted 2021-12-29 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Knee Arthroplasty (Active Comparator): Surgical knee replacement using either total knee replacement (TKA) or unicompartmental knee replacement (UKA)
  Interventions: Procedure: Surgical knee arthroplasty
- Supervised weight loss program (Experimental): The supervised intensive dietary weight loss program with meal replacements
  Interventions: Behavioral: Supervised weight loss

INTERVENTIONS:
Procedure: Surgical knee arthroplasty — Surgery will be performed 3 months from inclusion in the trial (at week 13). The procedure and type of prosthesis and postoperative program will be at the discretion of the involved surgeon and the participating department.
  Post-surgical care and rehabilitation will follow current clinical standards.
  Arms: Knee Arthroplasty
Behavioral: Supervised weight loss — The supervised intensive dietary weight loss program will be initiated 3 months from inclusion in the trial (at week 13) and lasts for 12 weeks.
  The program includes full meal replacement by a standard liquid energy intake in a supervised dietary program. Participants will attend the nutrition department weekly. They will be weighed on a decimal scale, given nutritional and dietetic instructions by an experienced dietitian and formula diet products are handed in sessions of 1-2 h. The participants will be taught to make diet plans.
  Following the 12 weeks intensive dietary weight loss program participants will be scheduled for two booster follow-up sessions with a dietician at weeks 39 and 51.
  Arms: Supervised weight loss program

SUMMARY:
This study addresses this question by comparing two recommended and potentially competing strategies in the management of obese knee OA patients:

Strategy A. A 3-months waiting list followed by a 12-week Intensive supervised diet intervention; Strategy B. A 3-months waiting list followed by surgical knee arthroplasty including standard post-operative rehabilitation.

The primary outcome is taken at week 38 from inclusion (baseline) corresponding to 6 months after treatment start (either surgery or intensive diet program).

Outcomes are also taken at baseline, week 13 (before treatment start), week 26 (end of diet program), week 38 (primary endpoint), and week 64.

DETAILED DESCRIPTION:
This trial asks a previously unaddressed and important clinical question about management of knee osteoarthritis (OA) patients.

Current recommendations of management of knee OA highlight weight loss as first choice and weight loss is a potential principal intervention against knee OA as a co-morbidity to obesity.

Knee arthroplasty (KA) is an effective treatment of knee OA in patients with pain that limits the patient's ability to perform their normal daily activities. KA is considered a successful orthopedic procedure to alleviate knee pain and disability in end stage knee OA. The demand for KA is large and growing worldwide; in Denmark alone approximately 10,000 KA procedures are performed annually, which pose a substantial economic burden to the health care system. KA carries relatively low risk both in terms of systemic complications and suboptimal outcomes for the joint itself. KA is one of the most effective surgical procedures available with very few contraindications. As a result, the demand from patients for these treatments continues to rise along with the confidence of surgeons to offer KA to a wider range of patients in terms of age, disability and co-morbidities.

However, the quality of evidence for KA efficacy is low as very few randomized controlled trials (RCTs) exist - particularly with respect to comparative effectiveness. To inform decision making for obese individuals with knee OA, it is important to evaluate the comparative effectiveness of a weight loss intervention against KA. The present trial has been designed to compare the effectiveness of weight loss and KA in individuals with obesity and knee OA.

This study addresses this question by comparing two recommended and potentially competing strategies in the management of obese knee OA patients:

Strategy A. A 3-months waiting list followed by a 12-week Intensive supervised diet intervention; Strategy B. A 3-months waiting list followed by surgical knee arthroplasty including standard post-operative rehabilitation.

Although a trial to address this question is needed, so far this study has not been carried out, presumably because trials in routine clinical practice are quite expensive and health care professionals (HCPs) responsible for delivery of either strategy have little incentive to compare KA to less expensive, non-surgical therapies. Moreover, the Danish Health and Medicines Authority have not required such comparisons. Since the Danish healthcare system already provides KA at public hospitals, it appears that such settings are ideally suited to address this question and, in the process, help clinicians around the world make better judgments for their patients with OA.

The sparse comparative effectiveness evidence that could inform clinical decision making, combined with existing evidence from RCTs and observational studies on knee surgery and weight loss provide a clear-cut ethical and scientific justification for the trial described in this protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or more
2. A clinical and radiological diagnosis of knee OA
3. BMI ≥ 30 kg/m2
4. Motivated for weight loss as by the provided program
5. Signed informed consent.

Exclusion Criteria:

1. The scheduled surgery is for revision of an existing prosthesis
2. Planned surgery for more than one knee within the observation period
3. KA indication due to sequelae of fracture(s)
4. Injection of medication or substances in the target knee within 3 months prior to participation
5. Immuno-inflammatory arthritis as cause of the knee OA
6. Current systemic treatment with glucocorticoids equivalent to > 7.5 mg of prednisolone/day
7. Previous or planned obesity surgery
8. Inability to understand or read Danish incl. instructions and questionnaires
9. Any other condition or impairment that, in the opinion of the investigator (or his/her delegate), makes a potential participant unsuitable for participation or which obstruct participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2022-01-13 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2025-02-24 (Actual)

PRIMARY OUTCOMES:
The Oxford Knee Score | Week 38 from baseline
  The Oxford Knee Score (OKS) is a 12-item Patient Reported Outcome questionnaire developed specifically to assess the patient's perspective on the outcomes of KA with respect to combined pain and physical function. Standardized answer options are given (5 Likert boxes) and each question is assigned a score from 0 to 4. Thus, a total score is calculated that ranges from 0 and 48, with 48 indicating the best outcome. The OKS is short, practical, reliable, valid, and sensitive to clinically important changes over time.

SECONDARY OUTCOMES:
The EuroQoL Health outcome and quality of life questionnaire (EQ-5D-5L) | Week: 13, 26, 38 and 64 from baseline
  EQ-5D-5L is a standardized patient-reported instrument for use as a measure of health outcome and quality of life. EQ-5D-5L is designed for self-completion by respondents and is ideally suited for use in surveys.
  The EQ-5D-5L consists of a descriptive system and the EQ Visual Analogue scale (EQ VAS). The descriptive system comprises 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). Standardized answer options are given (5 Likert boxes) and each question is assigned a score from 1 to 3.
  A country-specific index score is calculated.
Proportion of participants with Metabolic syndrome | Week: 13, 26, 38 and 64 from baseline
  Metabolic Syndrome (MetS) is defined according to the Harmonized definition: MetS is present when three or more of the following conditions occur simultaneously:
  * Elevated waist circumference (≥94 cm in men and ≥80 cm for women)
  * Elevated triglycerides (drug treatment for elevated triglycerides is an alternate indicator) ≥150 mg/dL (1.7 mmol/L)
  * Reduced HDL-C (drug treatment for reduced HDL-C is an alternate indicator) <40 mg/dL (1.0 mmol/L) in males; <50 mg/dL (1.3 mmol/L) in females
  * Elevated blood pressure (antihypertensive drug treatment in a patient with a history of hypertension is an alternate indicator) Systolic ≥130 and/or diastolic ≥85 mm Hg
  * Elevated fasting glucose (drug treatment of elevated glucose is an alternate indicator) ≥100 mg/dL
Change in proportions of participants the use analgesics for knee OA pain. | Week: 13, 26, 38 and 64 from baseline
  At clinical outcome assessment visit, the participants will be interviewed by an investigator about their use of analgesics since last visit. The interview will be focused on intake of
  1. Paracetamol/acetaminophen
  2. NSAIDS
  3. Acetylic acids
  4. Opioids The use of these analgesics will be recorded as use/non-use
The 12 item short form of tge Knee injury and Osteoarthritis Outcome Score (KOOS-12) | Week: 13, 26, 38 and 64 from baseline
  KOOS-12 is a 12-item measure derived from the original 42-item Knee injury and Osteoarthritis Outcome Score. KOOS-12 provides scores for knee-specific Pain, Function and QOL, along with a summary measure of overall knee impact. KOOS-12.
  Each item is scored from 0 to 4, left to right, with 0 representing no knee problems and 4 representing extreme knee problems. The KOOS-12 Summary knee impact score is calculated as the average of the Pain, Function and QOL scores that are calculated on a 0-100 scale, where 0 is the worst possible and 100 is the best possible score.
Patient's global assessment of impact of the knee in daily life (PGA) | Week: 13, 26, 38 and 64 from baseline
  The participant's assessment (PGA) of the impact of their knee on everyday life is measured as the response to the question "Taking into account all the activities you have during your daily life, your level of pain, and your functional impairment, how much does your [left/right] knee impact your daily life?". A 100 mm visual analogue scale (VAS) will be used as assessment instrument with anchors: 0 = "No impact" and 100 = "Worst imaginable impact".
Timed up-and-go | Week: 13, 26, 38 and 64 from baseline
  The timed up-and-go test (TUG) is a physical performance test primarily measuring the participants' ability to turn whilst walking (ambulatory transitions).
  The TUG measures the time it takes a participant to rise from a standard armchair, walk as quickly, but as safely as possible, a distance of 3 m, turn, walk back to the chair and sit down. Usual footwear and regular walking aids are allowed and recorded. The fastest of two trials is recorded in seconds. The same chair is used for all tests in this trial.
Patient Acceptable Symptom State (PASS) | Week: 13, 26, 38 and 64 from baseline
  PASS is assessed as yes/no answer to the question: "Taking into account all the activities you have during your daily life, your level of pain, and also your functional impairment, do you consider that your current state is satisfactory?".
  Those who reply 'no' the PASS question will be asked to answer (yes/no) the following question: "Would you consider your current state as being so unsatisfactory that you think the treatment has failed?" Participants replying, 'yes' to this second question will be defined as experiencing 'treatment failure' (TF).
  Besides the above algorithm treatment failure (TF) is also reached for:
  1. Participants in the KA group that during the observation period undergo revision surgery, And,
  2. Patients in the intensive diet group that during the observation period chose to undergo knee surgery.
Proportion of patients who experience minimal important improvement | Week: 13, 26, 38 and 64 from baseline
  A global transition questionnaire in which patients are asked to rate how they experience their health status has changed since before a treatment.
  The participants answer the question "How do you experience your knee problems now compared to prior to your study participation? Predefined answers are provided with scores ranging from -3 (worsening) to 3 (improvement):
  * 3: Worse, an important deterioration
  * 2: Somewhat worse, but enough to be an important deterioration
  * 1: Very small change, not enough to be an important deterioration 0: About the same
    1. Very small change, not enough to be an important improvement
    2. Somewhat better, but enough to be an important improvement
    3. Better, an important improvement
  From the transition scores, a predefined cut-off to define participants who experience minimally important improvement is set to a score of at least 2.
Proportion of participants that meet the OMERACT-OARSI response criteria | Week: 13, 26, 38 and 64 from baseline
  Per the Outcome Measures in Rheumatology (OMERACT) and Osteoarthritis Research Society International (OARSI) - (OMERACT-OARSI) criteria, a participant is classified as a (positive) responder if at least one of the following two conditions is observed at the post-Baseline assessment:
  • In either KOOS-12 pain subscale or KOOS-12 function subscale, both a > 50% improvement from Baseline and an absolute change from Baseline of > 20 units (0-100 scale),
  OR Improvement in at least two of the following three:
  1. Improvement in KOOS-12 pain subscale of > 20% improvement from Baseline and an absolute change from Baseline of > 10 normalized points (0-100 scale)
  2. Improvement in KOOS-12 function subscale defined as > 20% improvement from Baseline and an absolute change from Baseline of > 10 normalized points (0-100 scale)
  3. Improvement in PGA defined as > 20% improvement from Baseline and an absolute change from Baseline of > 10 mm (0-100 mm scale)
Body weight | Week: 13, 26, 38 and 64 from baseline
  The participants body weight is measured using a calibrated digital scale. The measurement is taken in kilograms (kg) recorded with 1 decimal.

OTHER OUTCOMES:
Change in number of steps per day | baseline and week 13, 26, 38 and 64
  Measurement of step counts will be done using wrist-worn activity trackers designed to measure steps (step counter). The participants will be asked to wear the step counter on the non-dominant wrist continuously (24 hours/day) for a 7-day period.
Assessment of glycemic control by plasma levels of glucose | baseline and week 13, 26, 38 and 64
  Glucose will be measured from fasting blood samples
Assessment of glycemic control by plasma levels of glycated hemoglobin (glycohemoglobin, HbA1c) | baseline and week 13, 26, 38 and 64
  HbA1c will be measured from fasting blood samples
Plasma levels of total cholesterol, low-density lipoprotein (LDL) cholesterol, high-density lipoprotein (HDL) cholesterol, and triglycerides | baseline and week 13, 26, 38 and 64
  Plasma lipids will be measured from fasting blood samples
Systolic and diastolic blood pressure | baseline and week 13, 26, 38 and 64
  Systolic and diastolic blood pressures are measured using a standard blood pressure apparatus.
Fat mass and lean body mass | baseline and week 38 and 64
  Body composition as well as bone mineral measurements will be assessed via whole-body dual energy X-ray absorptiometry (DEXA) using a Norland scanner. From the same scan, the following parameters will be recorded; fat mass (kg), lean body mass (kg).
Brief Illness perception questionnaire (B-IPQ) | baseline and week 13, 26, 38 and 64
  Brief Illness perception questionnaire (B-IPQ) is a generic 8-item questionnaire developed to rapidly assess the cognitive and emotional representations in a variety of illnesses.
  Five of the items assess cognitive illness representations; two of the items assess emotional representations; and one item assesses illness comprehensibility.
  Each item is scored on a 4 point Likert scale (0-3) with higher scores indicating worse illness perception. No sum score is calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- The Parker Institute, Frederiksberg Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided